CLINICAL TRIAL: NCT00675415
Title: Does Capnography Prevent Hypoxemia During ERCP and EUS? A Randomized, Controlled Trial
Brief Title: Does Capnography Prevent Hypoxemia During Endoscopic Retrograde Cholangiopancreatography and Endoscopic Ultrasound?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, John Vargo, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB#06-681
Record Dates: First submitted 2008-03-30; First posted 2008-05-09 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Hypoxemia
Keywords: Hypoxemia; Capnography; Apnea; Sedation; ERCP; EUS
MeSH Terms: conditions — Hypoxia; Apnea | interventions — Capnography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capnography (Active Comparator): Capnography: Subjects randomized to capnography-titration arm: The endoscopy team would be made aware of the capnographic abnormalities as they arise.
  In this arm, the endoscopy team will have the graphic representation of respiratory activity (capnography) as well as end-epxiratory levels of carbon dioxide in addition to the normal physiologic monitoring portfolio of pulse oximetry, blood pressure and electrocradiography.
  This observation phase would take place for a baseline prior to sedation, during the administration of sedation as well as throughout the procedure. Monitoring for the study would stop upon completion of the endoscopic procedure.
  Interventions: Diagnostic Test: Capnography
- Standard Monitoring (No Intervention): Subjects randomized to capnography-blinded arm: In this arm, the endoscopy team will not have the graphic representation of respiratory activity (capnography) as well as end-expiratory levels of carbon dioxide available. Only a standard of care physiologic monitoring portfolio of pulse oximetry, blood pressure and electrocradiography at the disposal of the endoscopy team to titrate the sedative medications.

INTERVENTIONS:
Diagnostic Test: Capnography — Capnography: Passive measurement of carbon dioxide via a special bite block which allows graphic assessment of the subject's respiratory activity
  Other Names: Oridion Capnomater and CapnoBiteBloc
  Arms: Capnography

SUMMARY:
Subjects undergoing elective ERCP and EUS will receive standard monitoring and sedation. In addition, capnography which measures carbon dioxide levels and can graphically assess respiratory activity will be used. Subjects will be randomized to either a capnography blinded or titration arm. In the capnography titration arm, the endoscopy team would be made aware of capnographic abnormalities as they arise throughout the procedure. In the capnography blinded arm, this information will not be available to the endoscopy team and represents standard of care. It is our hypothesis that using capnography can prevent low oxygen levels known as hypoxemia, during these procedures.

DETAILED DESCRIPTION:
Subjects undergoing elective ERCP and EUS will receive standard monitoring and sedation. In addition, capnography which measures carbon dioxide levels and can graphically assess respiratory activity will be used. Subjects will be randomized to either a capnography blinded or titration arm. In the capnography titration arm, the endoscopy team would be made aware of capnographic abnormalities as they arise throughout the procedure. In the capnography blinded arm, this information will not be available to the endoscopy team and represents standard of care. It is our hypothesis that using capnography can prevent low oxygen levels known as hypoxemia, during these procedures. The primary outcome of our study is the proportion of patients with hypoxemia in the two arms. Review of the literature indicates that the incidence of hypoxemia without supplemental oxygen varies from 30-70%. Our sample size calculation is based on a reduction of the hypoxemia incidence from 40% to 20%. Secondary outcomes will be the proportions of patients with oxygen requirements, major hypoxemia and apnea (lack of respiratory activity via capnography for at least 15 seconds) in the two arms. We will perform a univariable and multivariable analysis to determine the risk factors for apnea.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or greater
* Subjects undergoing elective ERCP and EUS
* ASA class 1-3
* Inpatient and outpatient
* Able to give informed consent

Exclusion Criteria:

* ASA Class 4 and 5
* Emergent procedures
* Procedures requiring MAC sedation
* Subjects unable to give informed consent
* Subjects on oxygen before procedure
* Subjects on CPAP/BiPAP
* Allergies to fentanyl/demerol/midazolam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Vargo, M.D., M.P.H., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qadeer MA, Vargo JJ, Dumot JA, Lopez R, Trolli PA, Stevens T, Parsi MA, Sanaka MR, Zuccaro G. Capnographic monitoring of respiratory activity improves safety of sedation for endoscopic cholangiopancreatography and ultrasonography. Gastroenterology. 2009 May;136(5):1568-76; quiz 1819-20. doi: 10.1053/j.gastro.2009.02.004. PMID 19422079

RESULTS

PARTICIPANT FLOW:
Groups:
- Capnography: Capnography: Subjects randomized to capnography-titration arm: The endoscopy team would be made aware of the capnographic abnormalities as they arise.
  In this arm, the endoscopy team will have the graphic representation of respiratory activity (capnography) as well as end-epxiratory levels of carbon dioxide in addition to the normal physiologic monitoring portfolio of pulse oximetry, blood pressure and electrocradiography.
  This observation phase would take place for a baseline prior to sedation, during the administration of sedation as well as throughout the procedure. Monitoring for the study would stop upon completion of the endoscopic procedure.
  Capnography: Capnography: Passive measurement of carbon dioxide via a special bite block which allows graphic assessment of the subject's respiratory activity
Period: Overall Study
Arm/Group | Capnography | Standard Monitoring
Started | 132 | 131
Completed | 124 | 123
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capnography | Standard Monitoring | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (14.4) | 60.6 (14.3) | 60.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 61 | 124
  Male | 61 | 62 | 123
Region of Enrollment [Number; unit: participants]
  United States | 124 | 123 | 247

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Hypoxemia During Endoscopy
Description: Hypoxemia was defined as oxygen saturation less than 90 percent for at least 15 seconds.
Time Frame: Continuously Assessed during a single endoscopic procedure, typically about 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Capnography | Standard Monitoring
Number analyzed (Participants) | 124 | 123
Participants | 57 | 85

2. Secondary Outcome: Proportion of Participants Requiring Supplemental Oxygen
Time Frame: Continuously measured during endoscopy, typically about 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Capnography | Standard Monitoring
Number analyzed (Participants) | 124 | 123
Participants | 65 | 82

3. Secondary Outcome: Proportion of Participants Experiencing Severe Hypoxemia
Time Frame: Continuously measured during endoscopy, typically about 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Capnography | Standard Monitoring
Number analyzed (Participants) | 124 | 123
Participants | 19 | 38

4. Secondary Outcome: Proportion of Participants Experiencing Apnea
Time Frame: Continuously measured during endoscopy, typically about 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Capnography | Standard Monitoring
Number analyzed (Participants) | 124 | 123
Participants | 51 | 77

ADVERSE EVENTS:
Time Frame: Measured continuously during each participant's endoscopic procedure, typically about two hours
Description: Capnography Monitoring system provides continuous measurement of breathing, pulse, and oxygen saturation information.
Arm/Group | Capnography | Standard Monitoring
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/123
Other Adverse Events (participants affected / at risk) | 101/124 | 95/123
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capnography (N=124) | Standard Monitoring (N=123)
Abnormal Breathing (Respiratory, thoracic and mediastinal disorders) | 101 | 95
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 57 | 85
Hypotension (Blood and lymphatic system disorders) | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes